## **Title Page**

#### **Protocol Title:**

Collection of Serum Samples From Children 6 Months to < 9 Years of Age Who Received Fluzone<sup>®</sup> Quadrivalent and Adults ≥ 65 Years of Age Who Received Fluzone<sup>®</sup> High-Dose Quadrivalent, Influenza Vaccines, 2020–2021 Formulations

**Study Code:** GRC00101

**Protocol Version Number: 1.0** 

Amendment Number: Not Applicable

Compound: Fluzone® Quadrivalent and Fluzone® High-Dose Quadrivalent Influenza Vaccines

(2020–2021 Formulations)

**Study Phase: IV** 

#### **Short Title:**

Annual Study for Collection of Serum Samples in Children and Older Adults Receiving the 2020–2021 Formulations of Fluzone Quadrivalent Vaccine and Fluzone High-Dose Quadrivalent Vaccine, Respectively

#### **Sponsor Name and Legal Registered Address:**

Sanofi Pasteur Inc.

Discovery Drive, Swiftwater, PA 18370-0187, USA

**Manufacturer:** Same as Sponsor

#### Regulatory Agency Identifier Numbers:

BB-IND: 4518

WHO UTN: U1111-1238-1821 NCT04551677

**Approval Date: 29 June 2020** 

#### Medical Monitor Name and Contact Information are provided in the Operating Guidelines.

The study centers, the Investigators at each center, and the Coordinating Investigator are listed in a separate document.

#### **Document History**

Not applicable as this is the first version of the protocol.

## **Table of Contents**

| List of | Tables | 6 |
|---|---|---|
| List of | Figures | 7 |
| 1 | Protocol Summary | 8 |
| 1.1 | Synopsis | 8 |
| 1.2 | Schema | 10 |
| 1.3 | Schedule of Activities (SoA) | 11 |
| 2 | Introduction | 15 |
| 2.1 | Study Rationale | 15 |
| 2.2<br>2.2.1<br>2.2.2<br>2.2.3<br>2.2.4 | Background Epidemiology Prevention and Control of Infection Among Humans The Advisory Committee on Immunization Practices Recommendations Background of the Investigational Product | 17<br>18<br>19 |
| 2.3<br>2.3.1<br>2.3.2<br>2.3.3 | Benefit/Risk Assessment Risks from Study Participation Benefits from Study Participation Overall Benefit-Risk Conclusion | 20<br>25 |
| 3 | Objectives and Endpoints | 25 |
| 4 | Study Design | 26 |
| 4.1 | Overall Design | 26 |
| 4.2 | Scientific Rationale for Study Design | 27 |
| 4.3 | Justification for Dose | 28 |
| 4.4 | End of Study Definition | 28 |
| 5 | Study Population | 28 |
| 5.1 | Inclusion Criteria | 28 |
| 5.2 | Exclusion Criteria | 29 |
| 5.3 | Lifestyle Considerations | 30 |
| 5.4 | Screen Failures | 30 |
| 6 | Study Intervention | 31 |

| 6.1 | Study Interventions Administered | 31 |
|---|---|---|
| 6.2 | Preparation/Handling/Storage/Accountability | 32 |
| 6.3<br>6.3.1<br>6.3.2 | Measures to Minimize Bias: Randomization and Blinding | 33 |
| 6.4 | Study Intervention Compliance | 33 |
| 6.5<br>6.5.1 | Concomitant Therapy | |
| 6.6 | Dose Modification | 34 |
| 6.7 | Intervention After the End of the Study | 35 |
| 7 | Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal | 35 |
| 7.1<br>7.1.1<br>7.1.2 | Discontinuation of Study Intervention | 35 |
| 7.2 | Participant Discontinuation/Withdrawal from the Study | 36 |
| 7.3 | Lost to Follow-up | 36 |
| 8 | Study Assessments and Procedures | 37 |
| 8.1<br>8.1.1<br>8.1.2 | Efficacy and Immunogenicity Assessments Efficacy Assessments Immunogenicity Assessments | 37 |
| 8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4 | Safety Assessments Medical History Physical Examinations Vital Signs Clinical Safety Laboratory Assessments | 38<br>38 |
| 8.3<br>8.3.1<br>8.3.2<br>8.3.3<br>8.3.4<br>8.3.5<br>8.3.6 | Adverse Events and Serious Adverse Events Time Period and Frequency for Collecting AE and SAE Information. Method of Detecting SAEs/AESIs Follow-up of SAEs and AESIs Regulatory Reporting Requirements for SAEs Pregnancy Adverse Events of Special Interest | 39<br>40<br>40 |
| 8.4 | Treatment of Overdose | |
| 8.5 | Pharmacokinetics | 41 |
| 8.6 | Pharmacodynamics | 41 |
| 8.7 | Genetics | 41 |

| 8.8 | Biomarkers | 41 |
|---|---|---|
| 8.9 | Immunogenicity Assessments | 41 |
| 8.10 | Health Economics or Medical Resource Utilization and Health Economics | 41 |
| 9 | Statistical Considerations | 42 |
| 9.1 | Statistical Hypotheses | 42 |
| 9.2 | Sample Size Determination | 42 |
| 9.3 | Populations for Analyses | 42 |
| 9.4 | Statistical Analyses | 42 |
| 9.4.1 | General Considerations. | |
| 9.4.2 | Primary Endpoint(s) | 42 |
| 9.4.3 | Secondary Endpoint(s) | 42 |
| 9.4.4 | Observational Endpoint(s) | 43 |
| 9.4.5 | Other Safety Analyse(s) | 43 |
| 9.4.6 | Other Analyse(s) | 43 |
| 9.5 | Interim Analyses | 43 |
| 9.6 | Data Monitoring Committee (DMC) | 43 |
| 10 | <b>Supporting Documentation and Operational Considerations</b> | 44 |
| 10.1 | Appendix: Regulatory, Ethical, and Study Oversight Considerations | 44 |
| 10.1.1 | Regulatory and Ethical Considerations | |
| 10.1.2 | Financial Disclosure | 44 |
| 10.1.3 | Informed Consent Process | 45 |
| 10.1.4 | Data Protection and Future Use of Stored Samples | 45 |
| 10.1.5 | Committees Structure | |
| 10.1.6 | Dissemination of Clinical Study Data | |
| 10.1.7 | Data Quality Assurance | |
| 10.1.8 | Source Documents | |
| 10.1.9 | Study and Site Start and Closure | |
| 10.1.10 | Publication Policy | 49 |
| 10.2 | Appendix: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting | 50 |
| 10.2.1 | Definition of AE | |
| 10.2.1 | Definition of SAE | |
| 10.2.2 | Recording and Follow-Up of AE and/or SAE | |
| 10.2.3 | Reporting of SAEs | |
| 10.2.5 | Assessment of Intensity | |
| 10.2.5.1 | • | |
| 10.3 | Appendix: Risk-based Approach | 56 |
| 10.4 | Appendix: Abbreviations | 57 |

| 10.5 | References | 58 |
|------|------------------------|----|
| 11 | Sponsor Signature Page | 61 |

## **List of Tables**

| Table 1.1: Schedule of Activities 1 | 12 |
|-------------------------------------------------------------------------|----|
| Table 1.2: Schedule of Activities 2 | 14 |
| Table 2.1: Potential Risks of Clinical Significance and Risk Management | 21 |
| Table 3.1: Objectives and Endpoints | 26 |
| Table 4.1: Overall Design | 27 |
| Table 6.1: Identity of Study Interventions | 31 |

## **List of Figures**

| Figure 1.1 – | - Graphical Study | Design for | Participants | 6 Months t | o < 9 Years | s of Age | 1 |
|---|---|---|---|---|---|---|---|
| Figure 1.2 – | - Graphical Study | Design for | Participants | > 65 Years | of Age | | 11 |

## **Protocol Summary**

#### 1.1 Synopsis

#### **Protocol Title:**

Collection of Serum Samples From Children 6 Months to < 9 Years of Age Who Received Fluzone<sup>®</sup> Quadrivalent and Adults ≥ 65 Years of Age Who Received Fluzone<sup>®</sup> High-Dose Quadrivalent, Influenza Vaccines, 2020–2021 Formulations

#### **Short Title:**

Annual Study for Collection of Serum Samples in Children and Older Adults Receiving the 2020–2021 Formulations of Fluzone Quadrivalent Vaccine and Fluzone High-Dose Quadrivalent Vaccine, Respectively

#### **Rationale:**

The aim of Study GRC00101 is to obtain serum samples for submission to the Center for Biologics Evaluation and Research (CBER) to aid in the influenza vaccine strain selection process. Children 6 months to < 9 years of age will receive the 2020–2021 formulation of Fluzone Quadrivalent vaccine and adults  $\ge 65$  years of age will receive the 2020–2021 formulation of Fluzone High-Dose Quadrivalent vaccine.

Serum samples from participants will be supplied to CBER after the completion of this study (i.e., after the last participant completes the last study visit). In turn, CBER will distribute the serum samples to the Centers for Disease Control and Prevention (CDC) and other World Health Organization (WHO)-collaborating laboratories for evaluation against circulating influenza viral strains. It is expected that the immunologic and surveillance data will be presented at WHO meetings where the vaccine strain selections will be made for the Southern and Northern hemispheres and at the Food and Drug Administration (FDA) Vaccines and Related Biological Products Advisory Committee meeting for selection of strains for influenza vaccines, including those to be distributed in the United States.

No early safety data review is planned for this study.

## **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To provide serum samples (collected from participants before vaccination [Blood Sample 1] and after final vaccination [Blood Sample 2]) to CBER for further analysis by the WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines. In addition, serum samples from adult participants may be further analyzed by the Sponsor to assess breadth of immune response induced by the study vaccines. | There are no endpoints for this objective. |

## **Overall Design:**

| Type of design | Parallel, multi-center |
|---|---|
| Phase | IV |
| Control Method | None |
| Study Population | Children 6 months to < 9 years of age<br>Adults ≥ 65 years of age |
| Countries | United States |
| Level and method of blinding | None (Open label) |
| Study intervention assignment method | Participants will not be randomized. |

**Disclosure Statement**: This is a parallel group serum collection study with 3 arms and no blinding.

## **Number of Participants:**

A total of 90 participants are expected to be enrolled. See Section 9.2.

#### **Intervention Groups and Duration:**

Each participant will be assigned to a vaccine group based on the participant's age at the time of enrollment.

- Group 1: Children 6 to < 36 months of age assigned to receive a 0.5-mL dose of Fluzone Quadrivalent vaccine (30 participants planned)
- Group 2: Children 3 to < 9 years of age assigned to receive a 0.5-mL dose of Fluzone Quadrivalent vaccine (30 participants planned)
- Group 3: Adults ≥ 65 years of age assigned to receive a 0.7-mL dose of Fluzone High-Dose Ouadrivalent vaccine (30 participants planned)

An approximately equal number of participants from each group will be enrolled at each site.

Participants will receive an intramuscular (IM) injection at Visit 1. For participants 6 months to < 9 years of age for whom 2 doses of influenza vaccine are recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second IM injection of Fluzone Quadrivalent vaccine will be administered at Visit 2 (28 [window, 28–35] days after Visit 1).

The duration of each subject's participation is as follows:

- Participants 6 months to < 9 years of age: 28 (window, 28–35) days following the last dose of influenza vaccine, including serious adverse event (SAE)/adverse event of special interest (AESI) follow-up. No additional safety follow-up beyond Visit 2 (for participants receiving 1 dose) or Visit 3 (for participants receiving 2 doses) is planned.</li>
- Participants ≥ 65 years of age: 21 (window, 21–28) days after vaccination, including SAE/AESI follow-up. No additional safety follow-up beyond Visit 2 is planned.

**Data Monitoring Committee: No** 

#### 1.2 Schema

The graphical designs of GRC00101 study are presented in Figure 1.1 and Figure 1.2.

Figure 1.1 – Graphical Study Design for Participants 6 Months to < 9 Years of Age



BL: blood sample VAC: vaccination

Figure 1.2 – Graphical Study Design for Participants ≥ 65 Years of Age



BL: blood sample VAC : vaccination

## 1.3 Schedule of Activities (SoA)

Visits procedures are detailed in the Operating Guidelines.

Participants receiving 2 doses of study vaccine, as per Advisory Committee on Immunization Practices (ACIP) guidance

Participants receiving 1 dose of study vaccine

**Table 1.1: Schedule of Activities 1** 

# For Participants 6 Months to < 9 Years of Age: Phase IV Study, 2 or 3 Visits, 1 or 2 Vaccinations, 1 or 2 Telephone Calls, 2 Blood Samples, 1 or 2 Months Duration Per Participant

| | All Participants | | | Participants<br>Receiving 1 Dose of<br>Influenza Vaccine | Participants Receiving 2 Doses of Influenza<br>Vaccine | | |
|---|---|---|---|---|---|---|---|
| Visit/Contact | Collection | Visit 1 | Telephone<br>Contact | Visit 2 | Visit 2 | Telephone<br>Contact | Visit 3 |
| Study timelines (days) | of information | Day 01 | Visit 1<br>+ 21 days | Visit 1 + 28 days | Visit 1<br>+ 28 days | Visit 2<br>+ 21 days<br>+ 19 to 23 days | Visit 2<br>+ 28 days |
| Time windows (days) | in the CRB | - | + 19 to 23 days | + 28 to 35 days | + 28 to 35<br>days | | + 28 to 35 days |
| Visit procedures: | | | | | | | |
| Informed consent/assent <sup>a</sup> | X | X | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | |
| Collection of demographic data | X | X | | | | | |
| Collection of medical history | X | X | | | | | |
| Influenza vaccination history | X | X | | | | | |
| History-directed physical examination | | X | | | X | | |
| Pre-vaccination temperature <sup>b</sup> | X | X | | | X | | |
| Review contraindications for vaccination | X | | | | X | | |
| Allocation of participant number | X | X | | | | | |
| Blood sampling (BL) <sup>c</sup> | X | BL1 | | BL2 | | | BL2 |
| Vaccination <sup>d</sup> | X | X | | | X | | |
| Immediate surveillance (20 minutes) | X | X | | | X | | |
| Diary card (DC) provided | | DC1 | | | DC2 | | |
| Telephone contacte | | | X | | | X | <u> </u> |

| | All Participants | | | Participants<br>Receiving 1 Dose of<br>Influenza Vaccine | Participants Receiving 2 Doses of Influenza<br>Vaccine | | of Influenza |
|---|---|---|---|---|---|---|---|
| Visit/Contact | Collection | Visit 1 | Telephone<br>Contact | Visit 2 | Visit 2 | Telephone<br>Contact | Visit 3 |
| Study timelines (days) | of information | Day 01 | Visit 1<br>+ 21 days | Visit 1 + 28 days | Visit 1<br>+ 28 days | Visit 2<br>+ 21 days | Visit 2<br>+ 28 days |
| Time windows (days) | in the CRB | | + 28 to 35 days | + 28 to 35 days | + 19 to 23 days | + 28 to 35<br>days | |
| Diary card reviewed | | | | DC1 | DC1 | | DC2 |
| Diary card collected | | | | DC1 | DC1 | | DC2 |
| Interim history | X | | | X | X | | X |
| Reporting medical events to allow<br>for the collection of SAEs and<br>AESIs | X | To be reported throughout the study period | | | | | |
| Collection of reportable concomitant medications | X | X | | X | X | | X |
| End of Active Phase participation record <sup>f</sup> | X | | | X | | | X |

AESI: adverse event of special interest; CRB: case report book; SAE: serious adverse event

- <sup>a</sup> Informed consent form will be signed and dated by parent(s) or guardian(s) for participants 6 months to < 9 years of age and assent form will be signed and dated by participants 7 to < 9 years of age.
- b The preferred route for this study is rectal for participants 6 to < 36 months of age, and oral for participants 3 to < 9 years of age. The axillary route may be used when a rectal or oral temperature cannot be obtained.
- <sup>c</sup> A blood sample, approximately 5 mL, will be collected from all participants at Visit 1, prior to vaccination, and at either Visit 2 (for participants receiving 1 influenza vaccine dose) or at Visit 3 (for participants receiving 2 influenza vaccine doses).
- d One or 2 doses of influenza vaccine will be administered according to the Advisory Committee on Immunization Practices guidance in effect during the study. If 2 doses of influenza vaccine are indicated, 1 dose will be administered during Visit 1 and the second dose will be administered approximately 28 days later during Visit 2.
- The participant's parent/guardian will be contacted by telephone 21 (window, 19–23) days after vaccination as a reminder to notify the site immediately if a serious medical event (e.g., hospital visit) occurs and to complete the diary card and to bring it with them to the next visit.
- The End of Active Phase participation record will be completed at Visit 2 for participants receiving 1 dose of influenza vaccine or at Visit 3 for participants receiving 2 doses of influenza vaccine. In case of participant discontinuation at a visit, the entire visit will be completed.

**Table 1.2: Schedule of Activities 2** 

## For Participants ≥ 65 Years of Age: 2 Visits, 1 Vaccination, 1 Telephone Call, 2 Blood Samples, 21 Days Duration Per Participant

| Visit/Contact | Collection | Visit 1 | Telephone<br>Contact | Visit 2 |
|---|---|---|---|---|
| Study timelines (days) | of<br>information<br>in the CRB | Day 01 | Visit 1 + 14 days | Visit 1 + 21<br>days |
| Time windows (days) | in the CKD | - | + 12 to 16 days | + 21 to 28 days |
| Visit procedures: | | | | |
| Informed consent | X | X | | |
| Inclusion/exclusion criteria | X | X | | |
| Collection of demographic data | X | X | | |
| Collection of medical history | X | X | | |
| Influenza vaccination history (previous season) | X | X | | |
| History-directed physical examination | | X | | |
| Pre-vaccination temperature <sup>a</sup> | X | X | | |
| Allocation of participant number | X | X | | |
| Blood sampling (BL) <sup>b</sup> | X | BL1 | | BL2 |
| Vaccination | X | X | | |
| Immediate surveillance (20 minutes) | X | X | | |
| Diary card provided | | X | | |
| Telephone contact <sup>c</sup> | | | X | |
| Diary card reviewed and collected | | | | X |
| Reporting of medical events to allow for the collection of SAEs, including AESIs | X | To be 1 | reported throughout th | e study period |
| Collection of reportable concomitant medications | X | X | | X |
| End of Active Phase participation record <sup>d</sup> | X | | | X |

AESI: adverse event of special interest; CRB: case report book; SAE: serious adverse event

- <sup>a</sup> The preferred route for this study for participants  $\geq$  65 years of age is oral.
- <sup>b</sup> A blood sample, approximately 20 mL, will be collected at Visit 1 and Visit 2.
- <sup>c</sup> Participants will be contacted by telephone 14 (window, 12–16) days after vaccination as a reminder to notify the site immediately if a serious medical event (e.g., hospital visit) occurs and to complete the diary card and to bring it with them to Visit 2.
- d In case of participant discontinuation at a visit, the entire visit will be completed.

#### 2 Introduction

## 2.1 Study Rationale

The aim of Study GRC00101 is to obtain serum samples for submission to CBER to aid in the influenza vaccine strain selection process. Children 6 months to < 9 years of age will receive the 2020–2021 formulation of Fluzone Quadrivalent vaccine and adults  $\ge 65$  years of age will receive the 2020–2021 formulation of Fluzone High-Dose Quadrivalent vaccine.

Serum samples from participants will be supplied to CBER after the completion of this study (i.e., after the last participant completes the last study visit). In turn, CBER will distribute the serum samples to the CDC and other WHO-collaborating laboratories for evaluation against circulating influenza viral strains. It is expected that the immunologic and surveillance data will be presented at WHO meetings where the vaccine strain selections will be made for the Southern and Northern hemispheres and at the FDA Vaccines and Related Biological Products Advisory Committee meeting for selection of strains for influenza vaccines, including those to be distributed in the United States.

No early safety data review is planned for this study.

#### 2.2 Background

This is a study using the 2020–2021 formulations of quadrivalent inactivated influenza vaccine (Fluzone Quadrivalent, Influenza Vaccine) and high-dose quadrivalent inactivated influenza vaccine (Fluzone High-Dose Quadrivalent, Influenza Vaccine).

Influenza viruses types A and B belong to the genus *Orthomyxoviridae* and are characterized as enveloped, negative-strand, segmented ribonucleic acid (RNA) viruses. The viral envelope contains 2 virus-coded glycoprotein spikes, the hemagglutinin (HA) and neuraminidase (NA) proteins, which are key antigens in the host response to influenza virus in both natural infection and vaccination. A third protein, M2, is a minor envelope component of the A-strain viruses (1).

Influenza is transmitted through inhalation of virus-containing droplets from infected individuals. The incubation period is usually 1 to 2 days (2). The virus multiplies in the ciliated columnar epithelium of the upper and lower respiratory tract, causing cellular necrosis and sloughing (1). Virus shedding typically begins just before illness onset (within 24 hours), rapidly peaks, and remains elevated for 1 to 2 days before rapidly declining to low levels. Usually, virus shedding lasts a total of 5 to 10 days (2).

There is considerable variation in the severity of illness in different individuals, partly due to age, general health, and immune status relative to previous influenza infections and vaccination. The classic symptoms include rapid onset (12 hours or less) of malaise, fever, myalgia, headache, and a non-productive cough or sore throat. Most symptoms last several days, but malaise and cough may last for a week or more (2). Complications of influenza include primary viral pneumonia,

secondary bacterial pneumonia, and exacerbation of underlying medical conditions such as chronic obstructive pulmonary disease and congestive heart failure.

While influenza affects all age groups, the elderly, children younger than 5 years of age, and persons with underlying health problems are amongst those at increased risk for complications. Members of high-risk groups who become ill with influenza are more likely than the general population to require hospitalization. Among infants and younger children, estimated rates of influenza-associated hospitalization are substantially higher than among older children and are similar to rates for other groups considered at higher risk for influenza-related complications, including persons  $\geq 65$  years of age who are at increased risk due to immunosenescence and adults 50-64 years of age and older who are at increased risk because they are likely to have chronic medical conditions that could lead to severe influenza illness (3).

Antigenic variation is an important feature of the influenza virus. The viral HA and NA surface antigens are subject to continuous and sequential evolution within immune or partially immune populations. Antigenic drift results from mutation(s) affecting the RNA segment coding for either HA or NA, but more commonly HA. As a result, there is alteration in protein structure involving 1 or a few amino acids, resulting in minor changes in antigenicity. Antigenic variants within a subtype (e.g., H1 or H3) emerge and through natural selection gradually become the more predominant circulating virus strain, while the preceding antigenic variant is suppressed by specific immunity in the population. In contrast to antigenic drift, antigenic shift represents the emergence of completely new subtypes, typically through gene reassortment with other circulating strains and acquisition of antigenically different gene sequences. Antigenic shift occurs at irregular intervals and may lead to pandemics (1) (2). While influenza B appears to be more genetically stable than influenza A, the dominant circulating B strain typically varies from season to season. For over a decade, both Yamagata and Victoria lineages have co-circulated during each season with varying prevalence (4). The large antigenic divergence between the 2 influenza B lineages limits antigenic cross-reactivity; therefore, immunity to 1 B lineage may not provide adequate protection against the other. Accordingly, switching from a trivalent vaccine to a quadrivalent vaccine is expected to prevent additional morbidity and mortality associated with mismatched influenza B strains that may occur with trivalent vaccines (4). With this in mind, Fluzone Quadrivalent vaccine and Fluzone High-Dose Quadrivalent vaccine were developed.

Vaccination with influenza vaccine is the primary method for preventing influenza and its severe complications. It has been shown to be effective in reducing influenza-associated morbidity and mortality in groups at increased risk for influenza-related complications such as infants and young children and persons 50 years of age and older. Of note, immune responses to the vaccine are lower in seniors than those in young healthy adults (3). Strategies to improve immune responses to the vaccine in the elderly population could provide substantial additional reductions in influenza-associated morbidity and mortality. One approach is to increase the dose of HA in inactivated vaccines. Previous studies evaluating the immune responses in terms of hemagglutination inhibition (HAI) antibodies with higher doses of HA per strain in different influenza vaccines support a dose-response effect (5).

Fluzone High-Dose Quadrivalent vaccine contains 60 µg HA per virus strain per dose, which is 4 times the amount of HA per strain per dose in Fluzone Quadrivalent vaccine. It was developed for use in the elderly to elicit enhanced immune responses against influenza through the use of

higher antigen content, with the goal of providing older adults with improved protection against the disease.

During this study, Fluzone Quadrivalent or Fluzone-High-Dose Quadrivalent vaccine will be administered according to the guidelines in the Prescribing Information and only to persons for whom the respective vaccine is indicated.

The objective of this study is to provide serum samples collected from children 6 months to < 9 years of age who receive Fluzone Quadrivalent vaccine and adults  $\ge 65$  years of age who receive Fluzone High-Dose Quadrivalent vaccine to CBER. The serum samples are used for further analysis by the WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines. In addition, serum samples from adult participants may be further analyzed by the Sponsor to assess breadth of immune response induced by the study vaccines.

#### 2.2.1 Epidemiology

Influenza is noted for occurring in epidemics. Typically, localized influenza epidemics begin abruptly, peak in 2 to 3 weeks, and last 5 to 6 weeks, although this can vary considerably by season (for example, the 2017–2018 season lasted 19 weeks (6)). The first sign of influenza in a community is usually reports of increased numbers of children with febrile respiratory illness, although a nursing home outbreak may be the first indication. Outbreaks in children are usually followed by the occurrence of influenza-like illness among adults. Following this is an increase in hospital admissions for pneumonia, exacerbation of chronic obstructive pulmonary disease, croup, and congestive heart failure. Increased absenteeism from school and the workplace occur as a late indicator. Finally, an increased number of deaths due to pneumonia and influenza are a highly specific indicator of influenza. However, due to the reporting delay and time course from infection to death, this indicator lags behind the others (2).

As with other viral respiratory infections, influenza is a seasonal disease. In the Northern Hemisphere, influenza is most likely to occur from November to April, and in the Southern Hemisphere from May to October. In tropical regions, it is more endemic, with periods of increased activity occurring more than once a year.

The public health impact of influenza is dramatic. Annually, from the 2010–2011 through 2017–2018 influenza season in the United States (US), the CDC estimated that influenza resulted in 9.3–49.0 million illnesses, 140,000–960,000 hospitalizations, and 12,000–79,000 deaths (7). Estimated annual overall hospitalizations and deaths attributable to influenza during this period in the United States were higher compared to historical data, with annual estimated hospitalizations ranging from approximately 55,000 to 431,000 per season (mean: 226,000) from 1979–1980 through 2000–2001 and deaths ranging from 3,000 to 49,000 each season from 1976–1977 through 2006–2007 (8) (9). During the 2010–2011 through 2017–2018 influenza seasons, annual estimates for influenza-related hospitalizations and deaths were highest (45%–72% and 69%–89% of overall estimates, respectively) among adults  $\geq$  65 years of age (10). During the 2017–2018 season, rates of hospitalization in all age groups were the highest seasonal rates seen since hospital-based surveillance was expanded in 2005 to include all ages, with an estimated 11.5 million cases of influenza in children, 30 million cases of influenza in adults 18–64 years of age, and more than 7.3 million cases in adults  $\geq$  65 years of age (11).

In the United States, death associated with laboratory-confirmed influenza virus infection among children < 18 years of age has been a nationally reportable condition since 2004. Since reporting began, the total number of influenza-associated deaths among children during 1 season has ranged from 37 (during the 2011–2012 season) to 186 (during the 2017–2018 season, as of April 19, 2019); this excludes the 2009 pandemic, when 358 pediatric deaths from 15 April 2009 through 2 October 2010 were reported to the CDC (12). During the 2009 pandemic, the majority of children who died had 1 or more underlying medical conditions previously associated with conferring a greater risk for influenza complications (13). During the 2017–2018 season, approximately 80% of the deaths occurred in children who had not received the 2017–2018 influenza vaccine (12).

Based on current understanding, the epidemiology of influenza B is characterized by major epidemics every 2–4 years. It causes infections in all age groups, including children, young adults, and the elderly. While influenza affects all age groups, young children remain at increased risk for complications and are more likely than the general population to require hospitalization. Influenza B has been associated with myalgia, myositis, pneumonia, and leukopenia in children (14) (15) (16). Influenza B infection in older adults leads to excess mortality in some annual epidemics. Across all ages, the burden of disease from influenza B is less than that from A/H3N2 but greater than that from A/H1N1. Overall, it is a significant cause of absenteeism, clinic visits, hospitalizations, and deaths (4).

#### 2.2.2 Prevention and Control of Infection Among Humans

Currently, the most effective measure for reducing the impact of influenza is to vaccinate persons at risk each year before the onset of the influenza season, especially persons at high risk for influenza-related complications. The ACIP of the CDC recommends that all eligible persons 6 months of age and older receive annual vaccination against influenza (3).

Influenza vaccine has been effective in reducing influenza-related morbidity and mortality. The effectiveness of the influenza vaccine in preventing or attenuating influenza illness depends in part on the age and immune competence of the vaccine recipient and on the similarity between the virus strains present in the vaccine and those circulating in the community. Most vaccinated children and young adults develop high post-vaccination HAI antibody titers. These antibodies are protective against illness caused by strains similar to those in the vaccine or the related variants that may emerge during outbreak periods. Elderly persons and persons with certain chronic diseases may develop lower post-vaccination antibody titers than healthy young adults and thus may remain susceptible to influenza-related upper respiratory infections. However, even if such older persons develop influenza illness despite vaccination, the vaccine can be effective in preventing lower-respiratory tract involvement or other secondary complications, thereby reducing the risk of hospitalization and death (3).

Annually, from the 2011–2012 through 2018–2019 influenza seasons in the United States, overall vaccine effectiveness ranged from 19% to 52%, for children 6 months to < 9 years of age it ranged from 25% to 68%, and for adults  $\ge 65$  years of age it ranged from 17% to 50% (17). The

a Preliminary estimates for 2018–2019.

CDC estimated that influenza vaccination prevented 11% of influenza-related hospitalizations during the  $2018-2019^b$  season and averted 2625 influenza-associated deaths among adults  $\geq 65$  years of age. In this same period, for persons < 18 years of age, an estimated 144 influenza-associated deaths were averted (18).

#### 2.2.3 The Advisory Committee on Immunization Practices Recommendations

Because children 6 to < 24 months of age are at substantially increased risk for influenza-related hospitalizations, and children 24 through 59 months of age are at increased risk for influenza-related clinic and emergency department visits, the ACIP recommends annual vaccination of all eligible children in these age groups. In recent years, the ACIP further expanded the age groups targeted for vaccination, and now recommends that all eligible persons 6 months of age and older receive annual influenza vaccination (3). The ACIP continues to emphasize the importance of vaccinating persons  $\ge$  6 months of age who have high-risk medical conditions (3).

If a child 6 months to < 9 years of age is receiving influenza vaccine for the first time, based on ACIP recommendations, 2 doses of influenza vaccine should be administered 4 weeks apart during the current season. This recommendation is based on studies demonstrating that vaccine effectiveness is lower among children who have never received influenza vaccine previously or who received only 1 dose in their first year of vaccination than it is among those children who received 2 doses in their first year of being vaccinated. Children 6 months to < 9 years of age who are adequately primed, based on influenza vaccination history, should receive 1 dose during the current season as per ACIP recommendations (3).

#### 2.2.4 Background of the Investigational Product

#### **Vaccine Testing and Release**

Before being released for clinical use, the 2020–2021 formulations of Fluzone Quadrivalent and Fluzone High-Dose Quadrivalent vaccines will have passed all approved release-testing requirements.

#### **Previous Clinical Experience: Fluzone Vaccine**

Fluzone vaccine was licensed in the United States in 1947 as a whole-virus preparation and it has been available since 1980 as a split-virus preparation. Numerous clinical trials have demonstrated its safety, immunogenicity, and effectiveness. Clinical trials, in which Fluzone vaccine was used as a comparator, have also demonstrated the safety and immunogenicity, and/or effectiveness of Fluzone vaccines.

#### Fluzone Quadrivalent Vaccine

In pre-licensure studies, Fluzone Quadrivalent vaccine, which contains 4 influenza strains (A/H1N1, A/H3N2, and 2 B strains [1 each from the Yamagata and Victoria lineages]), induced antibody responses that were comparable to those induced by trivalent Fluzone vaccine with respect to the strains contained in each vaccine. Pre-licensure studies also demonstrated that the safety profile of Fluzone Quadrivalent vaccine was similar to that of trivalent Fluzone vaccine.

-

b Latest data available.

Accordingly, Fluzone Quadrivalent vaccine offers the possibility of protecting against both B lineages simultaneously, without compromising vaccine safety (19) (20).

#### Fluzone High-Dose Vaccine

Fluzone High-Dose vaccine, a trivalent formulation with 60 µg HA per viral strain, has been shown in pre-licensure studies to elicit a higher immune response in the elderly than does Fluzone vaccine (15 µg HA per viral strain) (21) (22) (23). Solicited injection site and systemic reactions were reported more frequently with Fluzone High-Dose vaccine; however, these events were generally mild to moderate in intensity and transient. No safety concerns were identified. Moreover, a large-scale efficacy trial, which was conducted during 2 influenza seasons (2011–2012 and 2012–2013) and involved more than 30,000 persons, showed that Fluzone High-Dose vaccine was 24.2% more effective than Fluzone vaccine in preventing laboratory-confirmed symptomatic influenza in persons 65 years of age and older. The results of the study met the FDA-agreed criteria for demonstrating the superiority of Fluzone High-Dose vaccine compared with Fluzone vaccine for prevention of influenza disease in older adults (24).

#### Fluzone High-Dose Quadrivalent Vaccine

In a pre-licensure study (25), Fluzone High-Dose Quadrivalent vaccine, which contains 4 influenza strains (A/H1N1, A/H3N2, and 2 B strains [1 each from the Yamagata and Victoria lineages]), induced antibody responses that were comparable to those induced by trivalent Fluzone High-Dose vaccine with respect to the strains contained in each vaccine. The study also demonstrated that the safety profile of Fluzone High-Dose Quadrivalent vaccine was similar to that of Fluzone High-Dose vaccine.

The efficacy of Fluzone High-Dose is relevant to Fluzone High-Dose Quadrivalent since both vaccines are manufactured according to the same process and have overlapping compositions (26).

#### 2.3 Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks, reasonably expected adverse events (AEs), the potential risks, and uncertainties of Fluzone Quadrivalent vaccine and Fluzone High-Dose Quadrivalent vaccine may be found in the US Prescribing Information for the vaccine administered.

#### 2.3.1 Risks from Study Participation

The potential risks of clinical significance and risk management are summarized in Table 2.1.

Table 2.1: Potential Risks of Clinical Significance and Risk Management

| Potential Risk of Clinical<br>Significance | Summary of Data/<br>Rationale for Risk | Risk Management |
|---|---|---|
| Investigated Vaccine: Fluzone Quadrivalent Vaccine | | |
| Refer to the package insert for<br>more information regarding<br>potential risks | Identified and potential risks observed in clinical trials and/or post-marketing surveillance. | Exclusion/inclusion criteria take into account contraindications, warnings and precautions as defined in product label. |
| Injection site reactions | Most common injection site reactions in children 6 to < 36 months of age: pain or tenderness, erythema, and swelling | Injection site reactions are generally mild and usually resolve within 3 days |
| | Most common injection site reactions in children 3 to < 9 years of age: pain, erythema, and swelling | |
| Systemic reactions | Most common solicited systemic reactions in children 6 to < 36 months of age: irritability, abnormal crying, malaise, drowsiness, appetite loss, myalgia, vomiting, and fever Most common solicited systemic reactions in children 3 to < 9 years of age are: myalgia, malaise, and headache | Systemic findings most often affect persons who have had no prior exposure to the virus antigens in the vaccine (e.g., young children) (27). These reactions begin 6 to 12 hours after vaccination and usually resolve within 3 days. |
| Immediate allergic reactions | Immediate allergic reactions (e.g., hives, angioedema, allergic asthma, and systemic anaphylaxis) occur rarely after influenza vaccination. These reactions probably result from hypersensitivity to some vaccine component (28) (29) (30). | These types of reactions are exceedingly rare and would most likely occur in persons with a severe reaction to influenza vaccine in the past. Vaccine should not be administered to anyone who has had a severe allergic reaction to any component of the vaccine. |
| Guillain-Barré syndrome<br>(GBS) | Among persons who received the swine influenza vaccine in 1976, the rate of GBS that exceeded the background rate was < 10 cases/1,000,000 persons vaccinated. Evidence for a causal relationship of GBS with subsequent vaccines prepared from other influenza | Even if GBS were a true side effect of vaccination in the years after 1976, the estimated risk for GBS of approximately 1 additional case/1,000,000 persons vaccinated is substantially less than the risk for severe influenza, which |

| Potential Risk of Clinical<br>Significance | Summary of Data/<br>Rationale for Risk | Risk Management |
|---|---|---|
| | viruses is unclear. Obtaining strong epidemiologic evidence for such a possible limited increase in risk is difficult for such a rare condition as GBS, which has an annual incidence of 10–20 cases per 1,000,000 adults and stretches the limits of epidemiologic investigation (31). Investigations to date indicate that there is no substantial increase in GBS associated with influenza vaccines (other than the swine influenza vaccine in 1976) and that, if influenza vaccine does pose a risk, it is probably slightly more than 1 additional case per 1,000,000 persons vaccinated (32). | could be prevented by vaccination in all age groups. |
| Febrile Seizures | Analysis of reports collected by the Vaccine Adverse Events Reporting System during the 2010–2011 influenza season suggested an increased risk of febrile seizures among children younger than 2 years of age who received trivalent inactivated influenza vaccine (IIV3) (33). Using data collected through the CDC-sponsored Vaccine Safety Datalink (VSD) project, Tse et al (34) found an increased risk of fever-associated seizure occurring on the day of and 1 day after influenza vaccination in children 6 months through 4 years of age during the 2010–2011 influenza season. The risk was higher among children who received concomitant IIV3 vaccine and pneumococcal conjugate vaccine (PCV) 13-valent, and peaked at approximately age 16 months (44.9 cases per 100,000 doses). In a subsequent study that | The maximum estimated absolute excess risk due to concomitant administration of IIV3, PCV, and DTaP-containing vaccines compared with administration of these vaccines on separate days was 30 cases per 100,000 vaccinees. According to CDC, the risk of febrile seizure following influenza vaccination is small (36). |

| Potential Risk of Clinical<br>Significance | Summary of Data/<br>Rationale for Risk | Risk Management |
|---|---|---|
| Significance | over 5 influenza seasons (2005–2011), Duffy et al (35) reported that inactivated influenza vaccination in children 6–23 months of age was not an independent risk factor for febrile seizures, but revealed an increased risk of febrile seizure when influenza vaccine was given with either PCV or a diphtheria-tetanus-acellular-pertussis (DTaP)-containing vaccine. | |
| Investigated V | accine: Fluzone High-Dose Quadr | ivalent Vaccine |
| Refer to the package insert for more information regarding potential risks | Identified and potential risks observed in clinical trials and/or post-marketing surveillance. | Exclusion/inclusion criteria take into account contraindications, warnings and precautions as defined in product label. |
| Injection site reactions | Most common injection site reactions in adults ≥ 65 years of age: pain | Injection site reactions are generally mild and usually resolve within 3 days. |
| | | A Phase III study performed in persons ≥ 65 years of age demonstrated increased rates of solicited injection site reactions in participants receiving Fluzone High-Dose vaccine compared to persons receiving Fluzone vaccine but were typically mild and transient (23). |
| Systemic reactions | Most common solicited systemic reactions in adults ≥ 65 years of age: malaise, myalgia, and headache | A Phase III study performed in persons ≥ 65 years of age demonstrated increased rates of solicited systemic reactions in participants receiving Fluzone High-Dose vaccine compared to persons receiving Fluzone vaccine but were typically mild and transient (23). Placebocontrolled trials suggest that in elderly persons and in healthy young adults, split-virus influenza vaccine is not associated with higher rates of systemic symptoms when |

| Potential Risk of Clinical<br>Significance | Summary of Data/<br>Rationale for Risk | Risk Management |
|---|---|---|
| g | | compared with placebo injection (37). Safety monitoring of Fluzone High-Dose vaccine during the first year after licensure indicated a higher than expected number of gastrointestinal events compared with standard-dose vaccine, but otherwise no new safety concerns were identified (38). |
| Immediate allergic reactions | Immediate allergic reactions (e.g., hives, angioedema, allergic asthma, and systemic anaphylaxis) occur rarely after influenza vaccination. These reactions probably result from hypersensitivity to some vaccine component (28) (29) (30). | These types of reactions are exceedingly rare and would most likely occur in persons with a severe reaction to influenza vaccine in the past. Vaccine should not be administered to anyone who has had a severe allergic reaction to any component of the vaccine. |
| Guillain-Barré syndrome | Among persons who received the swine influenza vaccine in 1976, the rate of GBS that exceeded the background rate was < 10 cases/1,000,000 persons vaccinated. Evidence for a causal relationship of GBS with subsequent vaccines prepared from other influenza viruses is unclear. Obtaining strong epidemiologic evidence for such a possible limited increase in risk is difficult for such a rare condition as GBS, which has an annual incidence of 10–20 cases per 1,000,000 adults and stretches the limits of epidemiologic investigation (31). Investigations to date indicate that there is no substantial increase in GBS associated with influenza vaccines (other than the swine influenza vaccine in 1976) and that, if influenza vaccine does pose a risk, it is probably slightly more than | Even if GBS were a true side effect of vaccination in the years after 1976, the estimated risk for GBS of approximately 1 additional case/1,000,000 persons vaccinated is substantially less than the risk for severe influenza, which could be prevented by vaccination in all age groups and especially in persons ≥ 65 years of age and those who have medical indications for influenza vaccination. |

| Potential Risk of Clinical<br>Significance | Summary of Data/<br>Rationale for Risk | Risk Management |
|---|---|---|
| | 1 additional case per 1,000,000 persons vaccinated (32). | |
| | Study Procedures | |
| Vasovagal reactions (syncope),<br>or psychogenic reactions to<br>needle (vaccine injection or<br>blood sampling) | Anxiety-related reactions can occur following, or even before, any vaccination as a psychogenic response to the needle injection or blood draw, and may be accompanied by several neurological signs such as transient visual disturbance, paresthesia or seizure-like activity. | Observation period after vaccination for early detection and treatment. |

DTaP: diphtheria-tetanus-acellular-pertussis; GBS: Guillain-Barré syndrome; IIV3: trivalent inactivated influenza vaccine; PCV: pneumococcal conjugate vaccine; VSD: Vaccine Safety Datalink

#### 2.3.2 Benefits from Study Participation

The benefit to subjects participating in this study is potential protection from influenza disease following the receipt of the 2020–2021 formulation of Fluzone Quadrivalent or Fluzone High-Dose Quadrivalent vaccine.

#### 2.3.3 Overall Benefit-Risk Conclusion

Considering the measures taken to minimize risk to participants enrolled in this study, the potential risks that may result from study participation are balanced by the anticipated benefits that may be afforded to participants.

## **3** Objectives and Endpoints

The study objectives and the corresponding endpoints are described in Table 3.1.

**Table 3.1: Objectives and Endpoints** 

| Objectives | Endpoints |
|---|---|
| Primary | |
| • To provide serum samples (collected from participants before vaccination [Blood Sample 1] and after final vaccination [Blood Sample 2]) to CBER for further analysis by the WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines. In addition, serum samples from adult participants may be further analyzed by the Sponsor to assess breadth of immune response induced by the study vaccines. | There are no endpoints for this objective. |

## 4 Study Design

## 4.1 Overall Design

The design of the study is summarized in Table 4.1.

**Table 4.1: Overall Design** 

| Type of design | Parallel, multi-center |
|---|---|
| Phase | IV |
| Control method | None |
| St. L | Children 6 months to < 9 years of age |
| Study population | Adults ≥ 65 years of age |
| Level and method of blinding | None (Open label) |
| Study intervention assignment method | Participants will not be randomized. |
| Number of participants | 90 participants (30 from 6 months to < 36 months of age, 30 from 3 years to < 9 years of age, and 30 from 65 years and older) |
| Intervention groups | Each participant will be assigned to a vaccine group based on the participant's age at the time of enrollment to receive either 1 or 2 doses of Fluzone Quadrivalent vaccine as per ACIP guidance (participants 6 months to < 9 years of age) or 1 dose of Fluzone High-Dose Quadrivalent vaccine (participants ≥ 65 years of age). |
| Total duration of study participation | <ul> <li>Participants 6 months to &lt; 9 years of age: 28 (window, 28–35) days following the last dose of influenza vaccine (Visit 2 [for participants receiving 1 dose] or Visit 3 [for participants receiving 2 doses]).</li> <li>Participants ≥ 65 years of age: 21 (window, 21–28) days after vaccination.</li> </ul> |
| Countries | United States |
| Use of an Independent Data Monitoring<br>Committee, Dose Escalation<br>Committee, or similar review group | No |

## 4.2 Scientific Rationale for Study Design

Serum samples from participants will be supplied to CBER after the completion of this study (i.e., after the last participant completes the last study visit). In turn, CBER will distribute the serum samples to the CDC and other WHO-collaborating laboratories for evaluation against circulating influenza viral strains. It is expected that the immunologic and surveillance data will be presented at WHO meetings where the vaccine strain selections will be made for the Southern

and Northern hemispheres and at the FDA Vaccines and Related Biological Products Advisory Committee meeting for selection of strains for influenza vaccines, including those to be distributed in the United States.

#### 4.3 Justification for Dose

For participants 6 months to < 9 years of age: the vaccination schedule of 1 or 2 doses (as per ACIP guidance for children 6 months to < 9 years of age) for the influenza season is per standard practice for receipt of annual influenza vaccination.

For participants  $\geq$  65 years of age: The vaccination schedule of a single dose for the influenza season is per standard practice for receipt of annual influenza vaccination.

#### 4.4 End of Study Definition

A participant is considered to have completed the study if he/she has completed the last visit planned in the SoA.

The end of the study is defined as the date of the last visit of the last participant in the study.

However, for periodic safety reports, the study is considered completed when the clinical study report is finalized.

## 5 Study Population

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1 Inclusion Criteria

Participants are eligible for the study only if all of the following criteria are met:

- I01: Aged 6 months to < 9 years or  $\ge 65$  years of age on the day of first study vaccination (study product administration).
- I02: For participants 6 to < 12 months of age, born at full term of pregnancy ( $\ge$  37 weeks) and with a birth weight  $\ge$  5.5 lbs (2.5 kg).
- Informed consent form (ICF) has been signed and dated by participants  $\geq$  65 years of age.
- I04: Assent form has been signed and dated by participants 7 to < 9 years of age, and ICF has been signed and dated by parent(s) or guardian(s) for participants 6 months to < 9 years of age.

<sup>&</sup>lt;sup>c</sup> "6 months to < 9 years" means from the 6th month after birth to the day before the 9th year. "≥ 65 years" means from the day of the 65th birthday onwards.

I05: Participants and parent/guardian (of participants 6 months to < 9 years of age) are able to attend all scheduled visits and to comply with all study procedures.

#### 5.2 Exclusion Criteria

Participants are not eligible for the study if any of the following criteria are met:

- E01: Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Note: Participants may be considered eligible for enrollment if no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the participant would complete safety surveillance for the present study.
- E02: Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
- E03: Previous vaccination against influenza (in the 2020-2021 influenza season) with either study vaccine or another vaccine.
- E04: Receipt of immune globulins, blood, or blood-derived products in the 3 months preceding planned inclusion.
- E05: Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the 6 months preceding planned inclusion; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
- E06: Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to study vaccine or to a vaccine containing any of the same substances.
  - Note: The list of vaccine components is included in the Prescribing Information for each study vaccine.
- E07: Thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator.
- E08: Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
- E09: Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
- E10: Current alcohol abuse or drug addiction.

- E11: Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion.<sup>d</sup>
- E12: Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature ≥ 100.4°F [38.0°C]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
- E13: Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) or in-laws of the Investigator or employee with direct involvement in the proposed study.
- E14: History of serious adverse reaction to any influenza vaccine.
- E15: Personal history of Guillain-Barré syndrome (GBS).
- E16: Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
- E17: Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
- E18: Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

Note: Participants enrolled into this study will not be prohibited from donating blood for non-interventional studies or other purposes.

If the participant has a primary physician who is not the Investigator, the site should contact this physician with the participant's consent to inform him/her of the participant's participation in the study. In addition, the site should ask this primary physician to verify exclusion criteria relating to previous therapies, such as receipt of blood products or previous vaccines.

#### 5.3 Lifestyle Considerations

No other restrictions than the ones listed in the exclusion criteria or in the contraindications for subsequent vaccinations are required.

#### 5.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomly assigned to study intervention. Screening information is recorded in the source documents.

Individuals who do not meet the criteria for participation in this study (screen failure) can be rescreened.

Chronic illness may include, but is not limited to, cardiac disorders, renal disorders, autoimmune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases.

## **6** Study Intervention

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

## 6.1 Study Interventions Administered

Study interventions are described in Table 6.1.

**Table 6.1: Identity of Study Interventions** 

| Intervention Name | Fluzone Quadrivalent vaccine, No<br>Preservative (0.5-mL dose), 2020–<br>2021 formulation | Fluzone High-Dose Quadrivalent vaccine (0.7-mL dose), 2020–2021 formulation |
|---|---|---|
| Use | Other (as indicated in the prescribing material) | Other (as indicated in the prescribing material) |
| IMP and NIMP | IMP | IMP |
| Туре | Vaccine | Vaccine |
| Dose Formulation | Suspension for injection in a pre-filled syringe | Suspension for injection in a pre-filled syringe |
| Unit Dose<br>Strength(s) | <ul> <li>15 μg of HA of each of the following strains per dose:</li> <li>A/Guangdong-Maonan/SWL1536/2019 (H1N1)pdm09-like virus</li> <li>A/Hong Kong/2671/2019 (H3N2)-like virus</li> <li>B/Washington/02/2019 (B/Victoria lineage)-like virus</li> <li>B/Phuket/3073/2013 (B Yamagata lineage)-like virus</li> </ul> | <ul> <li>60 μg of HA of each of the following strains per dose:</li> <li>A/Guangdong- Maonan/SWL1536/2019 (H1N1)pdm09-like virus</li> <li>A/Hong Kong/2671/2019 (H3N2)- like virus</li> <li>B/Washington/02/2019 (B/Victoria lineage)-like virus</li> <li>B/Phuket/3073/2013 (B Yamagata lineage)-like virus</li> </ul> |

| Excipients/Diluent | Formaldehyde, egg protein, octylphenol ethoxylate (Triton X-100), sodium phosphate-buffered isotonic sodium chloride solution | Formaldehyde, egg protein, octylphenol ethoxylate (Triton X-100), sodium phosphate-buffered isotonic sodium chloride solution |
|---|---|---|
| Dosage Level | 0.5 mL per dose | 0.7 mL per dose |
| Number of Doses /<br>Dosing Interval | 1 or 2 doses 28 days apart for children aged 6 months to < 9 years (as per ACIP guidance) | 1 dose |
| Route of Administration | IM injection | IM injection |
| Site of<br>Administration | Anterolateral muscle of the thigh or the deltoid muscle | Deltoid muscle |
| Sourcing | Provided by the Sponsor | Provided by the Sponsor |
| Packaging and<br>Labeling | Fluzone Quadrivalent and Fluzone High-Dose Quadrivalent vaccines will be supplied with their manufacturer's commercial labeling and packaging. | |
| Current/Former<br>Name(s) or Alias(es) | Not applicable | Not applicable |
| <b>Batch Number</b> | TBD | TBD |

Note: Strains are based on WHO/FDA recommendations for the 2020-2021 NH influenza season

ACIP: Advisory Committee on Immunization Practices; FDA: Food and Drug Administration; HA: hemagglutinin;

IM: intramuscular; IMP: Investigational Medicinal Product; NH: Northern Hemisphere;

NIMP: Non Investigational Medicinal Product; TBD: to be determined; WHO: World Health Organization

## 6.2 Preparation/Handling/Storage/Accountability

Detailed guidance and information are provided in the Operating Guidelines.

- 1) The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- 2) Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.

- 3) The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).
- 4) Further guidance and information for the final disposition of unused study interventions are provided in the Operating Guidelines.

## 6.3 Measures to Minimize Bias: Randomization and Blinding

#### **6.3.1** Randomization and Allocation Procedures

Participants will not be randomized. Each participant will be assigned to a vaccine group based on the participant's age at the time of enrollment.

Participant numbers will be 12 digits long, with a 3-digit country identifier, a 4-digit study center identifier, and a 5-digit participant identifier. The 5-digit participant identifier will correspond to the chronological order of enrollment in the center. For example, Participant 840000100001 is the first participant enrolled in Center Number 1 (in the United States) and Participant 840000200002 is the second participant enrolled in Center Number 2 (in the Unites States).

Participant numbers should not be reassigned for any reason.

#### **6.3.2** Blinding and Code-breaking Procedures

This is an open-label study.

#### **6.4** Study Intervention Compliance

The following measures will ensure that the vaccine doses administered comply with those planned, and that any noncompliance is documented so that it can be accounted for in the data analyses:

- All vaccinations will be administered by qualified and trained study personnel
- The person in charge of study intervention management at the site will maintain accountability records of study intervention delivery to the study site, study intervention inventory at the site, dose(s) given to each participant, and unused or wasted doses

#### 6.5 Concomitant Therapy

At the time of enrollment, ongoing medications and other therapies (e.g., blood products) should be recorded in the source document as well as new medications prescribed for new medical conditions/AEs during study participation.

Documentation in the case report book (CRB) of ongoing concomitant medication(s) will be limited to specific categories of medication(s) of interest beginning on the day of first vaccination. This may include medications of interest that were started prior to the day of vaccination.

Reportable medications will be collected in the CRB from the day of each vaccination to the end of the follow-up period (i.e., from Visit 1 through Visit 2 for participants receiving 1 dose of study vaccine or from Visit 1 through Visit 3 for participants receiving 2 doses of study vaccine).

Reportable medications include medications that impact or may impact the consistency of the safety information collected after any vaccination and/or the immune response to vaccination. As Category 1 medications are NOT reportable for this study, there are 2 standard categories of reportable medications, defined as follows:

- Category 2: medications impacting or that may have an impact on the immune response
  (e.g., other vaccines, blood products, antibiotic classes that may interfere with bioassays
  used by the Global Clinical Immunology [GCI] department or other testing laboratories,
  systemic steroids/corticosteroids, immune-suppressors, immune-modulators with
  immunosuppressive properties, anti-proliferative drugs such as DNA synthesis inhibitors)
- Category 3: medications impacting or that may have an impact on both the safety and the immune response (e.g., systemic steroids/corticosteroids)

The information reported in the CRB for each reported medication will be limited to:

- Trade name
- Origin of prescription: prophylaxis Yes/No. Medication(s) prescribed for AE prophylaxis will be recorded in the Action Taken of the AE collection tables.
- Medication category (2 or 3)
- Start and stop dates

Dosage and administration route, homeopathic medication, topical and inhaled steroids, as well as topical, ophthalmic, and ear treatments will not be recorded.

Topical analgesics should not be applied at the site of vaccination; however, if they are applied inadvertently to the vaccination site, they should be recorded as a Category 3 medication.

Medications given in response to an AE will be captured in the "Action Taken" section of the AE case report form (CRF) only. No details will be recorded in the concomitant medication CRF unless the medication(s) received belongs to one of the pre-listed categories. Medications will not be coded.

#### 6.5.1 Rescue Medicine

Appropriate medical equipment and emergency medications, including epinephrine (1:1000), must be available on site in the event of an anaphylactic, vasovagal, or other immediate allergic reaction.

#### 6.6 Dose Modification

Not applicable.

#### 6.7 Intervention After the End of the Study

Not applicable.

# 7 Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

## 7.1 Discontinuation of Study Intervention

#### 7.1.1 Temporary Contraindications

Should a participant experience one of the conditions listed below, the Investigator will postpone further vaccination until the condition is resolved. Postponement must still be within the timeframe for vaccination indicated in the SoA.

TCI01: Febrile illness (temperature  $\geq 100.4^{\circ}F \geq 38.0^{\circ}C$ ) or moderate or severe acute illness /infection on the day of vaccination, according to Investigator judgment

#### 7.1.2 Definitive Contraindications

Participants will permanently discontinue (definitive discontinuation) study intervention for the reasons listed below. These participants must not receive any additional dose of study intervention but should continue to be followed for safety. Additional unscheduled visits may be performed for safety reasons and information will be reported in the source documents.

Should a participant experience 1 of the conditions listed below, the Investigator will discontinue vaccination:

- DCI01: An anaphylactic or other significant allergic reaction to the previous dose of vaccine
- DCI02: Receipt of any non-study vaccine (including a non-study dose of 2020–2021 influenza vaccine), immune globulins, blood, or blood-derived products between Visit 1 and Visit 2.
- DCI03: Bleeding disorder, receipt of anticoagulants, or thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator.
- DCI04: Development of any condition that in the opinion of the Investigator would pose a health risk to the participant or could interfere with the evaluation of the study vaccine (including GBS, clinically significant developmental delay, neurologic disorder, seizure disorder, human immunodeficiency virus infection, hepatitis B, or hepatitis C).
- DCI05: Development of immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy; or receipt of long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks).
- DCI06: Adverse events that are considered a contraindication for further participation in the study.

#### 7.2 Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons. This is expected to be uncommon.
- The reason for withdrawal should be clearly documented in the source documents and in the CRB: Adverse Event, Lost to Follow-up, Protocol Deviation, or Withdrawal by Participant or Parent/Guardian/Legally Acceptable Representative.
- The participant will be permanently discontinued both from the study intervention and from the study at that time.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws consent, he/she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.
- Withdrawn participants will not be replaced.

#### Follow-up of Discontinuations

For participants who have prematurely terminated the study, the site should attempt to contact them and complete all scheduled safety follow-ups, except if they specified that they do not want to be contacted again and it is documented in the source document. For participants where the reason for early termination is lost to follow-up, the site will not attempt to obtain further safety information. See Section 7.3 for definition of "lost to follow-up".

## 7.3 Lost to Follow-up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the site for a required study visit or cannot be contacted as planned in the SoA:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods), or at least to determine his/her health status while fully respecting his/her rights. These contact attempts should be documented in the participant's medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.
Discontinuation of specific sites or of the study as a whole are handled as part of Appendix 10.1.

# **8 Study Assessments and Procedures**

- Study procedures and their timing are summarized in the SoA. Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria. The investigator will maintain a screening log to
  record details of all participants screened and to confirm eligibility or record reasons for
  screening failure, as applicable. There are no screening criteria other than the inclusion
  and exclusion criteria.

Blood samples will be collected as described in the SoA tables (Section 1.3).

The maximum amount of blood collected from each participant over the duration of the study, including any extra assessments that may be required, will not exceed 10 mL for participants 6 months to < 9 years of age or 40 mL for participants  $\ge 65$  years of age. Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

Guidance and information for the sample collection, preparation, storage, and shipment are provided in the Operating Guidelines.

# 8.1 Efficacy and Immunogenicity Assessments

## **8.1.1** Efficacy Assessments

No clinical efficacy data will be obtained in the study.

## **8.1.2** Immunogenicity Assessments

No immunogenicity data will be obtained in the study.

## 8.2 Safety Assessments

This section presents safety assessments other than AEs, which are presented in Section 8.3.

Planned time points for all safety assessments are provided in the SoA tables (Section 1.3).

## 8.2.1 Medical History

Prior to enrollment, participants will be assessed for pre-existing conditions and illnesses, both past and ongoing. Any such conditions will be documented in the source document. Significant (clinically relevant) medical history (reported as diagnosis) including conditions/illnesses for which the participant is or has been followed by a physician or conditions/illnesses that could resume during the course of the study or lead to an SAE/AESI or to a repetitive outpatient care will be collected in the CRB.

## 8.2.2 Physical Examinations

At Visit 01, the Investigator or a delegate will perform a history-directed physical examination. Information will be recorded in the source document.

## 8.2.3 Vital Signs

Oral (participants 3 years to < 9 years and participants  $\ge$  65 years of age) or rectal (participants 6 months to < 36 months) pre-vaccination temperature will be systematically collected by the investigator on the source document. Tympanic, skin, and temporal artery thermometers must not be used.

## 8.2.4 Clinical Safety Laboratory Assessments

Not applicable.

#### **8.3** Adverse Events and Serious Adverse Events

The definitions of an AE, SAE, and the different categories of AEs can be found in Appendix 10.2.

Participants or parents/guardians (of participants 6 months to < 9 years of age) will be instructed to record information about any medical events that might represent SAEs or AESIs that may occur from Visit 1 through Visit 2 (Diary Card 1) for all participants and from Visit 2 through Visit 3 (Diary Card 2) for participants receiving 2 doses of study vaccine. Space will be provided in the diary card for this purpose.

AEs will be reported by the participants/participants' parents/guardians to the investigator, then by the investigator to the Sponsor.

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an SAE/AESI and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study (see Section 7).

#### 8.3.1 Time Period and Frequency for Collecting AE and SAE Information

#### Immediate Post-vaccination Observation Period

Participants will be kept under observation for 20 minutes after each vaccination to ensure their safety. Any SAEs/AESIs during this post-vaccination observation should be documented in the source document.

#### **AESIs**

Adverse events of special interest will be collected from Visit 1 to Visit 2 for participants receiving 1 dose of study vaccine, and from Visit 1 to Visit 3 for participants receiving 2 doses of study vaccine.

See Section 8.3.6 for the list of AESIs.

#### SAEs

Information on SAEs will be collected and assessed throughout the study, from Visit 1 to Visit 2 for participants receiving 1 dose of study vaccine, and from Visit 1 to Visit 3 for participants receiving 2 doses of study vaccine. However, before the first study intervention administration, only SAEs related to study procedures are to be collected.

Medical occurrences that begin before the start of study intervention but after obtaining informed consent will not be recorded on the AE section of the CRB.

All SAEs will be recorded and reported to the Sponsor or designee immediately and under no circumstance should this exceed 24 hours, as indicated in Appendix 10.2. The investigator will submit any updated SAE data to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AE or SAE after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the Sponsor.

## 8.3.2 Method of Detecting SAEs/AESIs

Individual diary cards, specifically designed for this study by the Sponsor and provided to the study sites, will be given to study participants for the recording of safety information. These diary cards will include free text to capture additional safety information or other relevant details.

At specified intervals, the Investigator or an authorized designee will interview the participants or participants' parents/guardians to collect the information recorded in the diary card, and will attempt to clarify anything that is incomplete or unclear. All clinical study information gathered by the study site will be reported electronically by the Investigator or authorized designee using a web-based CRB. Any information that was not documented in the diary card will first be captured in the source document and then reported electronically.

Care will be taken not to introduce bias when detecting SAEs/AESIs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about SAE occurrences.

## 8.3.3 Follow-up of SAEs and AESIs

Unless a participant/participant's parent guardian refuses further contact, each participant who experiences an SAE e/AESI during the study must be followed until the condition resolves, becomes stable, or becomes chronic (even after the end of the participant's participation in the study) if *either* of the following is true:

- The SAE/AESI is considered by the Investigator to be related to the study intervention administered
- The SAE/AESI caused the discontinuation of the participant from the study or from vaccination

The Investigator will inform the Sponsor of the date of final disappearance of the event or the date of "chronicity" establishment.

## 8.3.4 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of a SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The Sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The Sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, Institutional Review Boards (IRB)/Independent Ethics Committees (IEC), and investigators.
- For all studies except those investigating medical devices investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and Sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing a SAE or other specific safety information (e.g., summary or listing of SAEs) from the Sponsor will review and then file it and will notify the IRB/IEC, if appropriate according to local requirements.

## 8.3.5 Pregnancy

Not applicable as the study does not include women of childbearing potential.

<sup>&</sup>lt;sup>e</sup> The classification of an SAE is determined by the GPV Department and RMO(s) at Sanofi Pasteur. GPV: Global Pharmacovigilance; RMO: Responsible Medical Officer

## 8.3.6 Adverse Events of Special Interest

Adverse events of special interest will be captured as SAEs. These include new onset of GBS, encephalitis/myelitis (including transverse myelitis), neuritis (including Bell's palsy, optic neuritis, and brachial neuritis), thrombocytopenia, vasculitis, convulsions (including febrile convulsions [children only]), and anaphylaxis or other hypersensitivity/allergic reactions from Visit 1 through Visit 2 for participants receiving 1 dose of vaccine, or from Visit 1 through Visit 3 for participants receiving 2 doses of vaccine.

#### **8.4** Treatment of Overdose

Since the study intervention is administered by a health care professional, it is unlikely that overdose by injection occurs.

However, in the event of an overdose, the investigator should:

- 1) Contact the Medical Monitor immediately.
- 2) Closely monitor the participant for any AE/SAE.
- 3) Document the quantity of the excess of the overdose in the source documents.

#### 8.5 Pharmacokinetics

Pharmacokinetics parameters are not evaluated in this study.

## 8.6 Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

#### 8.7 Genetics

Genetics are not evaluated in this study.

#### 8.8 Biomarkers

Biomarkers are not evaluated in this study.

## 8.9 Immunogenicity Assessments

See Section 8.1.2.

## 8.10 Health Economics or Medical Resource Utilization and Health Economics

Medical Resource Utilization and Health Economics parameters are not evaluated in this study.

## 9 Statistical Considerations

# 9.1 Statistical Hypotheses

No hypotheses will be tested. Only descriptive statistical analyses will be conducted in this study.

## 9.2 Sample Size Determination

The study will enroll approximately 90 participants: approximately 30 participants 6 to < 36 months of age will be administered Fluzone Quadrivalent vaccine (Group 1), approximately 30 participants 3 to < 9 years of age will be administered Fluzone Quadrivalent vaccine (Group 2), and approximately 30 participants  $\ge$  65 years of age will be administered Fluzone High-Dose Quadrivalent vaccine (Group 3).

No study power calculation will be conducted for this study.

## 9.3 Populations for Analyses

The following population is defined:

| Population | Description |
|---|---|
| All Vaccinated Participants Population | Participants who have received at least 1 dose of the study vaccine. |

## 9.4 Statistical Analyses

No statistical analysis plan (SAP) will be written for this study. This section of the protocol will be followed to provide descriptive tables and listings of data.

#### 9.4.1 General Considerations

Summaries of baseline demographic characteristics of the study participants will be presented. The number of participants enrolled and their age at enrollment (mean, median, and minimum and maximum), sex, race, and ethnic origin will be summarized, along with the number and description of protocol deviations. Listings of participants by age group, sex, vaccine received, and history of vaccination in the previous season will be provided.

## 9.4.2 Primary Endpoint(s)

There are no primary endpoints for this study.

## 9.4.3 Secondary Endpoint(s)

There are no secondary endpoints for this study.

## 9.4.4 **Observational Endpoint(s)**

There are no observational endpoints for this study.

## 9.4.5 Other Safety Analyse(s)

Listings or tables of SAEs and AESIs will be provided.

## 9.4.6 Other Analyse(s)

Not applicable.

# 9.5 Interim Analyses

This study will not include an early safety data review. However, participant safety will be continuously monitored by the Sponsor's internal safety review committee which includes safety signal detection at any time during the study.

No analyses are planned to be performed prior to the formal completion of the study.

# 9.6 Data Monitoring Committee (DMC)

Not applicable.

# 10 Supporting Documentation and Operational Considerations

## 10.1 Appendix: Regulatory, Ethical, and Study Oversight Considerations

Note: The term "participant" is used throughout this protocol. However, the term "subject" will be used in the CRB in order to comply with the Clinical Data Interchange Standards Consortium (CDISC) requirements.

## **10.1.1** Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
  - Applicable International Council for Harmonisation (ICH) Good Clinical Practice (GCP)
     Guidelines
  - Applicable laws and regulations
- The protocol, protocol amendments, ICF, Investigator Brochure (IB), and other relevant documents (e.g., advertisements) must be submitted to an IRB/IEC by the investigator or the Sponsor (according to local regulations) and reviewed and approved by the IRB/IEC before the study is initiated
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants
- The investigator or the Sponsor (according to local regulations) will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
- The investigator will be responsible for providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

#### 10.1.2 Financial Disclosure

Information related to financial disclosure is described in the Investigator's contract.

#### 10.1.3 Informed Consent Process

- The investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants or their
  parents/guardians will be required to sign a statement of informed consent that meets the
  requirements of 21 CFR 50, local regulations, ICH guidelines, Health Insurance Portability
  and Accountability Act (HIPAA) requirements, where applicable, and the IRB/IEC or study
  center.
- In addition to the ICF that is signed by the participant or participant's parent/guardian, participants 7 to < 9 years of age will be asked to review and sign a study assent form.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- The actual ICF used at each center may differ, depending on local regulations and IEC/IRB requirements. However, all versions must contain the standard information found in the sample ICF provided by the Sponsor. Any change to the content of the ICF must be approved by the Sponsor and the IEC/IRB prior to the form being used.
- If new information becomes available that may be relevant to the participant's or parents'/guardians' willingness to continue participation in the study, this will be communicated to him/her in a timely manner. Such information will be provided via a revised ICF or an addendum to the original ICF (and assent form).
- Participants must be re-consented to the most current version of the ICF(s) and assent during their participation in the study.
- A copy of the ICF(s)/assent must be provided to the participant or the participant's legally authorized representative.

#### Recruitment Procedures

Participants may be recruited from the general population. The site will ensure that any advertisements used to recruit participants (informational brochures, parent letters, posters, and other advertisements) are submitted to Sanofi Pasteur prior to submission to the IRB(s) for approval.

#### 10.1.4 Data Protection and Future Use of Stored Samples

- All personal data collected related to participants, Investigators, or any person involved in the study, which may be included in the Sponsor's databases, shall be treated in compliance with all applicable laws and regulations including the Global Data Protection Regulation (GDPR).
   Data collected must be adequate, relevant and not excessive, in relation to the purposes for which they are collected. Each category of data must be properly justified and in line with the study objective.
- Participants race and ethnicity will be collected in this study because these data are required by regulatory agencies (e.g., on African-American population for the FDA in the United

- States or on Japanese population for the Pharmaceuticals and Medical Devices Agency in Japan).
- Participants will be assigned a unique identifier by the Sponsor. Any participant records or datasets that are transferred to the Sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred to the Sponsor.
- The participant must be informed that his/her personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant as described in the informed consent.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the Sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.
- When archiving or processing personal data pertaining to the Investigator and/or to the participants, the Sponsor shall take all appropriate measures to safeguard and prevent access to this data by any unauthorized third party.
- Participant data will be used for this study and in support of the whole drug development program for the Investigational Product, including negotiations with payers and publication of results.
- Any unused part of the serum samples will be securely stored at the Sanofi Pasteur serology laboratory (GCI) up to 25 years after the end of the study. These samples are being retained in long-term storage to support answers to regulatory questions related to the product's licensure and the potential revalidation of the study results.
  - In addition, participants/parents/guardians (of participants 6 months to < 9 years of age) will be asked to indicate in the ICF whether they will permit the future use of any unused stored serum samples for other tests. If they refuse permission, the samples will not be used for any testing other than that directly related to this study. If they agree to this use, they will not be paid for giving permission. Anonymity of samples will be ensured. The aim of any possible future research is unknown today, and may not be related to this particular study. It may be to improve the knowledge of vaccines or infectious diseases, or to improve existing tests or develop new tests to assess vaccines. Human genetic tests will never be performed on these samples without specific individual informed consent.

## 10.1.5 Committees Structure

This study will not include an early safety data review. However, participant safety will be continuously monitored by the Sponsor's internal safety review committee which includes safety signal detection at any time during the study.

#### 10.1.6 Dissemination of Clinical Study Data

Sanofi shares information about clinical trials and results on publicly accessible websites, based on company commitments, international and local legal and regulatory requirements, and other clinical trial disclosure commitments established by pharmaceutical industry associations. These

websites include clinicaltrials.gov, EU clinicaltrialregister (eu.ctr), and sanofi.com, as well as some national registries.

In addition, results from clinical trials in patients are required to be submitted to peer-reviewed journals following internal company review for accuracy, fair balance, and intellectual property. For those journals that request sharing of the analyzable data sets that are reported in the publication, interested researchers are directed to submit their request to clinical study data request.com.

Individual participant data and supporting clinical documents are available for request at clinical study data request.com. While making information available we continue to protect the privacy of participants in our clinical trials. Details on data sharing criteria and process for requesting access can be found at this web address: clinical study data request.com.

## **10.1.7** Data Quality Assurance

- All participant data relating to the study will be recorded on electronic CRB unless transmitted to the Sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRB.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the CRB.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- Monitoring details describing strategy (e.g., risk-based initiatives in operations and quality such as Risk Management and Mitigation Strategies and Analytical Risk-Based Monitoring), methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the Monitoring Plan.
- The Sponsor or designee is responsible for the data management of this study including quality checking of the data.
- The Sponsor assumes accountability for actions delegated to other individuals (e.g., Contract Research Organizations).
- Study monitors will perform ongoing source data verification to confirm that data entered into the CRB by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICFs, pertaining to the conduct of this study must
  be retained by the investigator for 25 years after the signature of the final study report unless
  local regulations or institutional policies require a longer retention period. No records may be
  destroyed during the retention period without the written approval of the Sponsor. No records
  may be transferred to another location or party without written notification to the Sponsor.

#### 10.1.8 Source Documents

"Source data" are the data contained in source documents. Source documents are original documents or certified copies, and include, but are not limited to, diary cards, medical and hospital records, screening logs, informed consent/assent forms, telephone contact logs, and worksheets.

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data entered in the CRB that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Detailed guidance and information are provided in the Operating Guidelines.

## 10.1.9 Study and Site Start and Closure

Details on which clinical supplies are provided by the Sponsor or the site are described in the Operating Guidelines.

The study start date is considered the date of the first visit planned in the SoA of the first participant.

The Sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the Sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been either destroyed or returned to the Sponsor, all samples are shipped to the appropriate laboratories, the center study-site has all the documents necessary for archiving and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the Sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study intervention development

If the study is prematurely terminated or suspended, the Sponsor shall promptly inform the Investigators, the IECs/IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The Investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

# 10.1.10 Publication Policy

Information related to publication policy is described in the Investigator's contract.

# 10.2 Appendix: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.2.1 Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

## **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.

- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### Other Definitions

#### Adverse Reaction:

All noxious and unintended responses to a study intervention related to any dose should be considered adverse reactions (AR).

(The phrase "responses to a study intervention" means that a causal relationship between a study intervention and an AE is at least a reasonable possibility)

#### Immediate Event/Reaction:

Immediate events are recorded to capture medically relevant unsolicited systemic AEs (including those related to the study intervention administered) that occur within the first 30 minutes after vaccination.

## Injection Site Reaction/Administration Site Reactions:

An injection/administration site reaction is an AR at and around the injection/administration site. Injection/administration site reactions are commonly inflammatory reactions. They are considered to be related to the study intervention administered.

#### Systemic AE/AR:

Systemic AEs are all AEs that are not injection or administration site reactions. They therefore include systemic manifestations such as headache, fever, as well as localized or topical manifestations that are not associated with the vaccination or administration site (e.g., erythema that is localized but that is not occurring at the injection site).

Systemic AEs assessed as related to study intervention are referred as systemic ARs.

## Adverse Event of Special Interest (AESI):

An adverse event of special interest (serious or non-serious) is one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the study Sponsor to other parties (e.g., regulators) might also be warranted.

#### Reactogenicity / Solicited Reactions

A solicited reaction is an "expected" AR ion (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB.

By definition, solicited reactions are considered as being related to the study intervention administered.

For injectable vaccines, solicited reactions can either be solicited injection/administration site reactions or solicited systemic reactions.

#### Unsolicited AE/AR

An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions, i.e., pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination. For example, varicella or a solicited term such as headache starting after the solicited observation period (headache starting on Day 10 post-vaccination in the case where headache occurring between the day of vaccination and the next 7 days is pre-listed in the protocol and CRB as a solicited reaction).

An unsolicited AR is an unsolicited AE that is considered related to study intervention. Unsolicited AEs includes both serious (SAEs) and non-serious unsolicited AEs.

#### 10.2.2 Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

## A SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

## b. Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

## c. Requires inpatient hospitalization or prolongation of existing hospitalization

- In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### d. Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and

accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

## e. Is a congenital anomaly/birth defect

#### f. Other important medical event

- Medical or scientific judgment should be exercised in deciding whether expedited reporting
  is appropriate in other situations such as important medical events that may not be
  immediately life-threatening or result in death or hospitalization but may jeopardize the
  health of the participant or may require intervention to prevent one of the other outcomes
  listed in the above definition. These important medical events should also usually be
  considered serious.
- Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse, new-onset diabetes or autoimmune disease.

**Note:** <u>Serious</u> and <u>severe</u> are not synonymous. The term <u>severe</u> is often used to describe the intensity of a specific event as corresponding to Grade 3. This is not the same as <u>serious</u>, which is based on participant / event outcome or action criteria usually associated with events that pose a threat to a participant's life or functioning.

## 10.2.3 Recording and Follow-Up of AE and/or SAE

#### **AE and SAE Recording**

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (e.g., hospital progress notes, laboratory reports, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE/SAE information in the CRB.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to the Sponsor in lieu of completion of the CRB pages.
- There may be instances when copies of medical records for certain cases are requested by the Sponsor. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to the Sponsor.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

## **Assessment of Causality**

By convention, all SAEs reported at the injection site are considered to be related to the study intervention and therefore are referred to as reactions and do not require the Investigator's opinion on relatedness.

- Causality of SAEs will be recorded as follows:
  - For SAEs/AESIs, relationship to study intervention will be assessed by both the Investigator and the Sponsor. Sponsor assessment is entered in the GPV database only.
  - For SAEs only, the causal relationship to study procedures (related/not related to study procedures) will be assessed by both the Investigator and the Sponsor. Sponsor assessment is entered in the GPV database only.
- The Investigator will assess the *causal relationship* between each SAE/AESI and the study intervention administered <sup>6</sup> as either *not related* or *related*, based on the following definitions:
  - Not related The SAE/AESI is clearly/most probably caused by other etiologies such as an underlying condition, therapeutic intervention, or concomitant therapy; or the delay between vaccination and the onset of the SAE is incompatible with a causal relationship; or the SAE/AESI started before the first vaccination (screening phase, if applicable)
  - Related There is a "reasonable possibility" that the SAE/AESI was caused by the study intervention administered, meaning that there is evidence or arguments to suggest a causal relationship
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the IB and/or Product Information, for marketed products, in his/her assessment.
- For each SAE/AESI, the investigator **must** document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE/AESI has occurred and the investigator has minimal information to include in the initial report to the Sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE/AESI data to the Sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send a SAE/AESI follow-up report with the updated causality assessment.

-

<sup>&</sup>lt;sup>6</sup> Study intervention administered can correspond to either the investigational product or other products when no investigational product is administered at the visit

• The causality assessment is one of the criteria used when determining regulatory reporting requirements.

## Follow-up of SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the Sponsor to elucidate the nature and/or causality of the SAE/AESI as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study or during a recognized follow-up period, when available the investigator will provide the Sponsor with a copy of any post-mortem findings including histopathology.
- New or updated information will be recorded in the originally completed CRB.
- The investigator will submit any updated SAE data to the Sponsor within 24 hours of receipt of the information.
- Serious adverse events/AESIs likely to be related to the study intervention, that persist at the end of the study will be followed up by the Investigator until their complete disappearance or the stabilization of the participant's condition. The Investigator will inform the Sponsor of the date of final disappearance of the event or the date of "chronicity" establishment.

#### 10.2.4 Reporting of SAEs

## SAE Reporting to the Sponsor via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to the Sponsor will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) in order to report the event within 24 hours. The site will enter the SAE data into the electronic system as soon as it becomes available.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section).
- Details regarding SAE reporting can be found in the Operating Guidelines.

## SAE Reporting to the Sponsor via Paper CRF

- The SAE paper CRF can be sent to the Sponsor by 1 of the following means:
- By fax, to the following number: 1-570-957-2782
- In PDF format to the following e-mail address, using a method of transmission that includes password protection: PV.outsourcing@sanofi.com
- By express mail, to the following address:
- Sanofi Pasteur, Inc.
   Reception & Triage Case Management
   Global Pharmacovigilance Department
   Discovery Drive, Swiftwater, PA 18370

## Safety Emergency Call

If, as per the Investigator's judgment, a participant experiences a medical emergency, the Investigator may contact the Sponsor's responsible medical officers (RMOs) for advice on how to address any study related medical question or problem. The RMOs will be available 24 hours a day, 7 days a week, as needed. Contact information for each of the RMOs is provided in the Operating Guidelines.

This process does not replace the need to report an SAE/AESI. The Investigator is still required to follow the protocol-defined process for reporting SAEs/AESIs to the Global Pharmacovigilance Department (please refer to Section 10.2.4).

#### 10.2.5 Assessment of Intensity

Not applicable.

#### **10.2.5.1** Tables for Clinical Abnormalities

Not applicable.

# 10.3 Appendix: Risk-based Approach

ICH E6-R2 guideline for GCP is introducing the « risk-based approach » concept which permits to focus efforts on what is critical for a study and most specifically on Critical Data and Critical Processes. Critical data and processes are defined for the study with associated risks in the Study Risk Management Plan.

## 10.4 Appendix: Abbreviations

ACIP Advisory Committee on Immunization Practices

AE Adverse Event

AESI Adverse Event of Special Interest

AR Adverse Reaction

CBER Center for Biologics Evaluation and Research
CDC Centers for Disease Control and Prevention

CRB Case Report Book
CRF Case Report Form

DTaP Diphtheria-Tetanus-Acellular-Pertussis

FDA Food and Drug Administration
GBS Guillain-Barré Syndrome
GCI Global Clinical Immunology
GCP Good Clinical Practice

GPV Global Pharmacovigilance Department

HA Hemagglutinin

HAI Hemagglutination Inhibition

IB Investigator Brochure
ICF Informed Consent Form

ICH International Council for Harmonisation

IEC Independent Ethics Committee

IM Intramuscular

IND Investigational New Drug (Application)

IRB Institutional Review Board

IIV3 Trivalent Inactivated Influenza vaccine

NA Neuraminidase

RMO Responsible Medical Officer

RNA Ribonucleic Acid
SAE Serious Adverse Event
SoA Schedule of Activities

US United States

VSD Vaccine Safety Datalink
WHO World Health Organization

#### 10.5 References

- 1. Fiore AE, Bridges CB, Katz JM, Cox NJ. Inactivated influenza vaccines. In: Plotkin SA, Orenstein WA, Offit PA, editors. Vaccines. 6th ed. Edinburgh, UK: Elsevier/Saunders; 2012. p. 257-93.
- 2. Treanor JT. Influenza viruses, including avian influenza and swine influenza. In: Mandell GL, Bennett JE, Dolin R, editors. Mandell, Douglas, and Bennett's Principles and Practice of Infectious Diseases. 7th ed. New York, NY: Churchill Livingstone; 2010. p. 2265-88.
- 3. Grohskopf LA, Sokolow LZ, Broder KR, Walter EB, Bresee JS, Fry AM, et al. Prevention and Control of Seasonal Influenza with Vaccines: Recommendations of the Advisory Committee on Immunization Practices United States, 2017-18 Influenza Season. MMWR Recomm Rep. 2017;66(2):1-20.
- 4. Belshe RB. The need for quadrivalent vaccine against seasonal influenza. Vaccine. 2010;28 Suppl 4:D45-53.
- 5. Monto AS, Ansaldi F, Aspinall R, McElhaney JE, Montaño LF, Nichol KL, et al. Influenza control in the 21st century: Optimizing protection of older adults. Vaccine. 2009;27(37):5043-53.
- 6. Centers for Disease Control and Prevention Website. Influenza (Flu) 2017-2018 2019 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/about/season/flu-season-2017-2018.htm#anchor 1534865788578.
- 7. Centers for Disease Control and Prevention Website. Burden of influenza. 2020 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/about/burden/index.html.
- 8. Thompson WW, Shay DK, Weintraub E, Brammer L, Bridges CB, Cox NJ, et al. Influenza-associated hospitalizations in the United States. JAMA. 2004;292(11):1333-40.
- 9. Centers for Disease Control and Prevention. Estimates of deaths associated with seasonal influenza --- United States, 1976-2007. MMWR Morb Mortal Wkly Rep. 2010;59(33):1057-62.
- 10. Centers for Disease Control and Prevention Website. Past seasons estimated influenza disease burden. 2020 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/about/burden/past-seasons.html.
- 11. Centers for Disease Control and Prevention Website. Estimated influenza illnesses, medical visits, hospitalizations, and deaths in the United States 2017-2018 influenza season. 2019 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/about/burden/2017-2018.htm.
- 12. Centers for Disease Control and Prevention Website. Summary of the 2017-2018 influenza season. 2019 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/about/season/flu-season-2017-2018.htm.
- 13. Centers for Disease Control and Prevention. Prevention and control of seasonal influenza with vaccines. Recommendations of the Advisory Committee on Immunization Practices--United States, 2013-2014. MMWR Recomm Rep. 2013;62(RR-07):1-43.

- 14. Hu JJ, Kao CL, Lee PI, Chen CM, Lee CY, Lu CY, et al. Clinical features of influenza A and B in children and association with myositis. J Microbiol Immunol Infect. 2004;37(2):95-8.
- 15. Hite LK, Glezen WP, Demmler GJ, Munoz FM. Medically attended pediatric influenza during the resurgence of the Victoria lineage of influenza B virus. Int J Infect Dis. 2007;11(1):40-7.
- 16. Glezen WP, Couch RB, Taber LH, Paredes A, Allison JE, Frank AL, et al. Epidemiologic observations of influenza B virus infections in Houston, Texas, 1976-1977. American journal of epidemiology. 1980;111(1):13-22.
- 17. Centers for Disease Control and Prevention Website. Past seasons vaccine effectiveness. 2020 [cited 2020 June 02]. Available from: https://www.cdc.gov/flu/vaccines-work/past-seasons-estimates.html.
- 18. Chung J, Rolfes M, Flannery B, Prasad P, O'Halloran A, Garg S, et al. Effects of Influenza Vaccination in the United States During the 2018–2019 Influenza Season. Clin Infect Dis. 2020.
- 19. Greenberg DP, Robertson CA, Landolfi VA, Bhaumik A, Senders SD, Decker MD. Safety and immunogenicity of an inactivated quadrivalent influenza vaccine in children 6 months through 8 years of age. Pediatr Infect Dis J. 2014;33(6):630-6.
- 20. Greenberg DP, Robertson CA, Noss MJ, Blatter MM, Biedenbender R, Decker MD. Safety and immunogenicity of a quadrivalent inactivated influenza vaccine compared to licensed trivalent inactivated influenza vaccines in adults. Vaccine. 2013;31(5):770-6.
- 21. Keitel WA, Atmar RL, Cate TR, Petersen NJ, Greenberg SB, Ruben F, et al. Safety of high doses of influenza vaccine and effect on antibody responses in elderly persons. Arch Intern Med. 2006;166(10):1121-7.
- 22. Couch RB, Winokur P, Brady R, Belshe R, Chen WH, Cate TR, et al. Safety and immunogenicity of a high dosage trivalent influenza vaccine among elderly subjects. Vaccine. 2007;25(44):7656-63.
- 23. Falsey AR, Treanor JJ, Tornieporth N, Capellan J, Gorse GJ. Randomized, double-blind controlled phase 3 trial comparing the immunogenicity of high-dose and standard-dose influenza vaccine in adults 65 years of age and older. J Infect Dis. 2009;200(2):172-80.
- 24. DiazGranados CA, Dunning AJ, Kimmel M, Kirby D, Treanor J, Collins A, et al. Efficacy of high-dose versus standard-dose influenza vaccine in older adults. N Engl J Med. 2014;371(7):635-45.
- 25. Chang LJ, Meng Y, Janosczyk H, Landolfi V, Talbot HK. Safety and immunogenicity of high-dose quadrivalent influenza vaccine in adults ≥65 years of age: A phase 3 randomized clinical trial. Vaccine. 2019;37(39):5825-34.
- 26. Fluzone High-Dose Quadrivant [Package Insert]. Swiftwater, PA: Sanofi Pasteur Inc.; 2019.
- 27. Fiore AE, Shay DK, Haber P, Iskander JK, Uyeki TM, Mootrey G, et al. Prevention and control of influenza. Recommendations of the Advisory Committee on Immunization Practices (ACIP), 2007. MMWR Recomm Rep. 2007;56(RR-6):1-54.

- 28. Centers for Disease Control and Prevention. Epidemiology and Prevention of Vaccine-Preventable Diseases. 13 ed. Hamborsky J, Kroger A, Wolfe S, editors: Washington D.C. Public Health Foundation; 2015.
- 29. Woo EJ. Allergic reactions after egg-free recombinant influenza vaccine: reports to the US Vaccine Adverse Event Reporting System. Clin Infect Dis. 2015;60(5):777-80.
- 30. Woo EJ, Moro PL, Cano M, Jankosky C. Postmarketing safety surveillance of trivalent recombinant influenza vaccine: Reports to the Vaccine Adverse Event Reporting System. Vaccine. 2017;35(42):5618-21.
- 31. Seneviratne U. Guillain-Barré syndrome. Postgrad Med J. 2000;76(902):774-82.
- 32. Salmon DA, Proschan M, Forshee R, Gargiullo P, Bleser W, Burwen DR, et al. Association between Guillain-Barré syndrome and influenza A (H1N1) 2009 monovalent inactivated vaccines in the USA: a meta-analysis. Lancet (London, England). 2013;381(9876):1461-8.
- 33. Leroy Z, Broder K, Menschik D, Shimabukuro T, Martin D. Febrile seizures after 2010-2011 influenza vaccine in young children, United States: a vaccine safety signal from the vaccine adverse event reporting system. Vaccine. 2012;30(11):2020-3.
- 34. Tse A, Tseng HF, Greene SK, Vellozzi C, Lee GM. Signal identification and evaluation for risk of febrile seizures in children following trivalent inactivated influenza vaccine in the Vaccine Safety Datalink Project, 2010-2011. Vaccine. 2012;30(11):2024-31.
- 35. Duffy J, Weintraub E, Hambidge SJ, Jackson LA, Kharbanda EO, Klein NP, et al. Febrile Seizure Risk After Vaccination in Children 6 to 23 Months. Pediatrics. 2016;138(1).
- 36. Centers for Disease Control and Prevention Website. Childhood Vaccines and Febrile Seizures 2020 [cited 2020 June 02]. Available from: https://www.cdc.gov/vaccinesafety/concerns/febrile-seizures.html.
- 37. Mitchell DK, Ruben FL, Gravenstein S. Immunogenicity and safety of inactivated influenza virus vaccine in young children in 2003-2004. Pediatr Infect Dis J. 2005;24(10):925-7.
- 38. Moro PL, Arana J, Cano M, Menschik D, Yue X, Lewis P, et al. Postlicensure safety surveillance for high-dose trivalent inactivated influenza vaccine in the Vaccine Adverse Event Reporting System, 1 July 2010-31 December 2010. Clin Infect Dis. 2012;54(11):1608-14.

| 11 | Sponsor | <b>Signature</b> | Page |
|----|---------|------------------|------|
|----|---------|------------------|------|

| Document Number | Version Number |
|-----------------|----------------|
| CLI_00310135 | 1.0 |
| Project Code | |
| Flu seasonal | |
| Arficact Name | |
| Protocol Body | |

| | Approver Name | Date<br>(Universal Time) | Reason for Signature |
|----------|---------------|--------------------------|----------------------|
| Approval | | | |